CLINICAL TRIAL: NCT01938027
Title: A Pilot Study for the Evaluation of the Safety and the Efficacy of Transanal Total Mesorectal Excision
Brief Title: The Evaluation of the Safety and the Efficacy of Transanal Total Mesorectal Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Jae Hwan Oh, Head of Center for Colorectal Cancer, National Cancer Center, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-TAME; NCC-1210170 (Other Grant/Funding Number: The National Cancer Center, South Korea)
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Neoplasms; Colorectal Neoplasms; transanal surgery
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transanal total mesorectal excision (Experimental): Laparoscopy-assisted transanal total mesorectal excision
  Interventions: Procedure: Transanal total mesorectal excision

INTERVENTIONS:
Procedure: Transanal total mesorectal excision — Laparoscopy-assisted transanal total mesorectal excision

SUMMARY:
The purpose of this study is evaluation of the safety and the efficacy of transanal total mesorectal excision.

DETAILED DESCRIPTION:
Subjects will have their rectal cancer removed using a technique combining surgery through the anus and standard laparoscopy. Transanal visualization will be using endoscopy. At the end of the procedure, the rectum will be removed though the anus or ileostomy formation site, the bowel will be re-connected to the anus, and a temporary diverting stoma will be created, which is standard of care following surgery for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* age: 20-80 years
* biopsy-proven adenocarcinoma of the rectum
* clinical staging, (T1 or T2 or T3) with N0M0
* Rectal cancer located 4-12 cm from the anal verge
* ECOG performance status 2 or less

Exclusion Criteria:

* Synchronous colon cancer or other malignancy
* Obstructing rectal cancer
* Pregnant or breast-feeding
* Receiving any other study agents
* Fecal incontinence
* History of prior colorectal cancer or inflammatory bowel disease
* BMI > 30
* T3 rectal cancer not treated preoperatively with full-course chemoradiation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Total Mesorectal Excision(TME) quality | 1-5 years
  The quality of the mesorectum was determined using pathology reports and scored using three grades:
  * Complete: intact mesorectum with only minor irregularities of a smooth mesorectal surface. No defect is deeper than 5 mm, and there is no coning toward the distal margin of the specimen. There is a smooth circumferential resection margin on slicing.
  * Nearly complete: moderate bulk to the mesorectum, but irregularity of the mesorectal surface. Moderate coning of the specimen is allowed. At no site is the muscularis propria visible, with the exception of the insertion of the levator muscles.
  * Incomplete: little bulk to mesorectum with defects down onto muscularis propria and/or very irregular circumferential resection margin.

SECONDARY OUTCOMES:
30-day postoperative complications, No. of harvested LN | 1-5 years

OTHER OUTCOMES:
Oncologic outcome(2-year local recurrence free survival, 5-year survival) | 1-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hwan Oh, MD, PHD, Principal Investigator — NCC,Korea
Locations (1):
- Jae Hwan Oh, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Oh JH, Park SC, Kim MJ, Park BK, Hyun JH, Chang HJ, Han KS, Sohn DK. Feasibility of transanal endoscopic total mesorectal excision for rectal cancer: results of a pilot study. Ann Surg Treat Res. 2016 Oct;91(4):187-194. doi: 10.4174/astr.2016.91.4.187. Epub 2016 Sep 30. PMID 27757396